CLINICAL TRIAL: NCT03380377
Title: A Phase I/II Trial to Evaluate the Safety and Tolerability of Clazakizumab (Anti-IL-6 Monoclonal) As an Agent to Eliminate Donor Specific HLA Antibodies and Improve Outcomes of Patients With Chronic & Active Antibody-Mediated Rejection Post-Kidney Transplantation
Brief Title: Clazakizumab for Chronic and Active Antibody Mediated Rejection Post-Kidney Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanley Jordan, MD (Other)
Responsible Party: Sponsor-Investigator, Stanley Jordan, MD, Director of the Kidney Transplant Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 134733
Record Dates: First submitted 2017-08-03; First posted 2017-12-21 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Antibody-mediated Rejection; Kidney Transplant; Complications; Transplant Glomerulopathy; Transplant Glomerulopathy - Late Form; Transplant Glomerulopathy - Early Form; Kidney Transplant Rejection
Keywords: kidney transplant; Chronic antibody mediated rejection; donor specific antibody
MeSH Terms: interventions — clazakizumab

STUDY DESIGN:
Intervention Model Description: All ten patients enrolled will receive study medication (Clazakizumab, Vitaeris, Inc, Vancouver, Canada, B.C)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clazakizumab (Anti-IL-6 Monoclonal) (Experimental): All ten patients will be receiving clazakizumab (Anti-IL-6 Monoclonal) monthly for six months. Then patients will be scheduled for six month protocol biopsy. If biopsy and all clinical labs show benefit or stability (up to PI discretion), patients will continue receiving clazakizumab monthly for another six months. All patients completing twelve doses of clazakizumab will be scheduled for a twelve month protocol biopsy and last study visit. If at the 6 month protocol biopsy, no improvement was seen, PI will have patient come for their last study visit on month 12 post enrollment.
  Interventions: Drug: Clazakizumab

INTERVENTIONS:
Drug: Clazakizumab — Clazakizumab 25 mg subcutaneous monthly x 6 doses (or max of 12 doses) will be given to patients who are enrolled in this clinical trial.

SUMMARY:
Antibody mediated rejection (ABMR) is a unique, significant and often severe form of allograft rejection. This single center, phase I/II, open label single-arm exploratory study focuses on enrolling ten patients with biopsy proven chronic antibody medicated rejection and/or donor specific antibody present at time of biopsy. Patients who qualify will be receiving clazakizumab (anti-IL6 monoclonal antibody) monthly x six doses. A protocol biopsy will be performed at 6 months and if improvement is seen, patients will continue another six doses for up to 12 months. For those completing 12 doses, there will be a 12 month protocol biopsy. For those who only received six doses, the next and last study visit will be at 12 months from enrollment. Total study duration is 12 months.

DETAILED DESCRIPTION:
This is a single center, Phase I/II, open label single-arm exploratory study. The trial will primarily examine the safety and tolerability of clazakizumab given after the diagnosis of cABMR in 10 subjects (15-75yrs) who exhibit DSAs to their donor. Patients entered will also have been diagnosed with cABMR + TG post-transplant based on Banff 2015 criteria. Patients are required to have a eGFR > 30 mL/min/1.73m2 as calculated by the MDRD equation (Schwartz equation will be used to estimate CrCl for patients under 18 years of age) at entry. All patients will be recruited from the renal transplant program at Cedars-Sinai Medical Center. Once cABMR is diagnosed, donor-specific anti-HLA antibodies will be assessed (DSA) which are associated with cABMR and/or graft loss. DSA will be detected using solid phase assay systems currently utilized at the Cedars-Sinai Medical Center HLA Laboratory (Dr. Xiaohai Zhang Director, Phone: 310-423-4979)41. These anti-HLA antibodies may result naturally or from previous pregnancy, transfusions, or prior transplants. Patients treated with clazakizumab for cABMR will have labs for DSAs, and other monitoring labs as well as immunologic studies as outlined. In addition to the standard post-transplant immunosuppressive protocol, patients with cABMR will receive clazakizumab 25mg SC given every 4 weeks (30 days) for a total of 6 doses. If no safety/tolerability/efficacy issues are observed after the initial dose, patients will continue the protocol as outlined. A protocol biopsy will be performed after the 6th and after the 12th doses of clazakizumab to assess the allograft for evidence of cABMR/ABMR, including C4d staining and TG using Banff 2015 criteria14. Banff scoring will be compared between the index and protocol biopsy after cessation of therapy. Patients who have evidence of persistent allograft dysfunction may have non-protocol biopsies for cause. After completion of the clazakizumab therapy, patients will be followed up to assess allograft function and ABMR episodes as well as DSAs. The protocol is summarized in figure 14 below. Monitoring of Treg, Th17, Tfh and plasmablast as well as IL-6, and CRP levels will be performed in the Transplant Immunology Lab at Cedars-Sinai Medical Center at select time points (Dr. Mieko Toyoda Director, Phone: 310-423-8282). confirmation) they will continue monthly clazakizumab for an additional 6 months and will have a second biopsy at 12 month protocol. Immunologic and viral monitoring labs will be performed as indicated.

The subjects will be followed to determine if the use of clazakizumab for treatment of cABMR in this high-risk transplant population is safe and without infectious risks. In addition, the investigators will determine the effects of clazakizumab treatment on renal biopsy assessments performed at 6 months. Assessments of renal function, donor specific antibody, and Banff 2015 biopsy scores will be evaluated at that time. If improvement or stabilization observed, clazakizumab will be resumed monthly x 6 doses (starting day 180 to day 330) and last study visit will be day 365 with biopsy. Study investigators will assess the transplanted patients to determine the number who sustain a viable and functioning kidney allograft as well. In the event a patient does not show improvement after receiving 6 doses of clazakizumab, no further treatment will be given and the patient will return at Day 365 for a final study visit. All subjects will be evaluated on an intent-to-treat basis. The subject accrual rate will be limited to no more than 1-2 subjects per month in the initial three months to assure safety to all subjects. Repeat laboratories will be performed at the completion of clazakizumab therapy to determine effect on levels and correlation with any potential events.

Long term dosing option at conclusion of 12 months (after Study Day 365 visit) will be available for those patients who complete the 12 month protocol. Patients may continue to receive clazakizumab 25 mg subQ every 8 weeks long term, per PI discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-75 years at the time of screening.
2. Biopsy proven cABMR with TG on biopsy as defined by Banff 2015 and DSA positive at time of biopsy
3. Subject/Parent/Guardian must be able to understand and provide informed consent.
4. Pneumococcal vaccinated
5. Negative tuberculin ppd result or negative Quantiferon TB gold

Exclusion Criteria:

1. Multi-organ transplant (e.g. kidney and pancreas)
2. eGFR < 30 mL/min/1.73m2
3. Advanced Transplant Glomerulopathy (CG3)
4. Previous allergic reactions to monoclonal antibodies.
5. Lactating or pregnant females.
6. Women of child-bearing age who are not willing or able to practice FDA-approved forms of contraception during study and for 5 months after last dose.
7. HIV-positive subjects.
8. Subjects who test positive for HBV by HBVeAg/DNA or HCV infection [positive Anti-HCV (EIA) and confirmatory HCV RIBA].
9. Subjects with latent or active TB. Subjects must have negative Quantiferon TB gold test result.
10. Recent recipients of any licensed or investigational live attenuated vaccine(s) within two months of the screening visit j) A significantly abnormal general serum screening lab result defined as a WBC < 3.0 X 103/ml, a Hgb < 8.0 g/dL, a platelet count < 100 X 103/ml, an SGOT or SGPT > 3X upper limit normal
11. Individuals deemed unable to comply with the protocol.
12. Subjects with active CMV or EBV infection as defined by CMV-specific serology (IgG or IgM) and confirmed by quantitative PCR with or without a compatible illness.
13. Use of investigational agents within 4 weeks of participation.
14. History or active Inflammatory Bowel Disease or Diverticular Disease or gastrointestinal perforation
15. Recent infection (within past 6 weeks of screening) requiring any antibiotic use (oral, parenteral or topical).
16. Present or previous (within 5 years) malignancy except for basal cell carcinoma, fully excised squamous cell carcinoma of the skin or non-recurrent (within 5 years) cervical carcinoma-in-situ.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center Comprehensive Transplant Center
Locations (1):
- Norko Ammerman, Los Angeles, California, United States

REFERENCES:
- [Background] Choi J, Aubert O, Vo A, Loupy A, Haas M, Puliyanda D, Kim I, Louie S, Kang A, Peng A, Kahwaji J, Reinsmoen N, Toyoda M, Jordan SC. Assessment of Tocilizumab (Anti-Interleukin-6 Receptor Monoclonal) as a Potential Treatment for Chronic Antibody-Mediated Rejection and Transplant Glomerulopathy in HLA-Sensitized Renal Allograft Recipients. Am J Transplant. 2017 Sep;17(9):2381-2389. doi: 10.1111/ajt.14228. Epub 2017 Mar 10. PMID 28199785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
Started | 10
Completed | 8
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 51 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73m2] | 38.11 (12.23)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Donor Specific Antibody (DSA) Elimination or Reduction Based on Luminex HLA Testing
Description: Did clazakizumab eliminate or weaken donor specific antibody (DSA) mean fluorescence intensity (MFI) intensities? HLA antibodies were detected by the single antigen bead-based assay (One lambda, Los Angeles, CA). Donor HLA-specific antibodies were assessed throughout clazakizumab treatment for the first year. Detection of DSAs were only reported with MFI >2500.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Number of Participants With Stabilization of Clinical Features of cABMR Via BANFF Biopsy Grading Criteria.
Description: Does clazakizumab help stabilize pathologic features of antibody mediated rejection at 6 month protocol biopsies? Protocol kidney allograft biopsies were performed at 6 months and compared to the baseline biopsy which was assessed for study inclusion. Biopsy specimens were analyzed according to Banff 2017 classification.
Time Frame: 6 months
Population: 9 of 10 patients underwent the 6 month protocol biopsy (One patient was withdrawn from study at 3 months and did not complete the 6 month biopsy)
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Stabilization in Estimated Glomerular Filtration Rate (eGFR)
Description: Serum creatinine (mg/dl) collected to calculate eGFR
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
Number analyzed (Participants) | 8
ml/min/1.73m2 | 41.6 (14.2)

4. Secondary Outcome: Incidence of Treatment-related Adverse Events
Description: Adverse event monitoring in our patient population; did patients have treatment related adverse events and if so, how many events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Clazakizumab (Anti-IL-6 Monoclonal)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazakizumab (Anti-IL-6 Monoclonal) (N=10)
Sepsis due to pyelonephritis (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazakizumab (Anti-IL-6 Monoclonal) (N=10)
EBV Viremia (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 2 (2)
Pyelonephritis (Renal and urinary disorders) | 3 (4)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
C difficile infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Cough and/or Cold (Infections and infestations) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Arm swelling/cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema/warts on hands (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent dizziness (General disorders) | 1 (1)
Edema (General disorders) | 3 (5)
Itching on legs (Skin and subcutaneous tissue disorders) | 1 (1)
Swollen hand after exercise (General disorders) | 1 (1)
Uric acid elevated/gout in big toe (Musculoskeletal and connective tissue disorders) | 1 (1)
Excision of skin cancer lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginitis (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Our phase 2 trial has several limitations, including the lack of a randomized controlled design with a placebo-treated control arm, a small sample size and variability among the participants at baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT03380377/Prot_000.pdf